CLINICAL TRIAL: NCT07039968
Title: Standard Dose Versus High Dose Stereotactic Spine Radiosurgery for Metastatic Spinal Neoplasms - SHINE: A Prospective Randomized Trial
Brief Title: Standard Dose Versus High Dose Stereotactic Spine Radiosurgery for Metastatic Spinal Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University Hospital, Yun-Lin Branch (Other); National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202503019RINA
Record Dates: First submitted 2025-06-16; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Spinal Neoplasms
Keywords: spine metastasis; stereotactic spine radiosurgery
MeSH Terms: conditions — Spinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dose Spine Stereotactic Radiosurgery (Active Comparator): Participants randomized to this arm will receive Spine Stereotactic Radiosurgery (SSRS) delivered at a dose of 16 Gray (Gy) in a single treatment session.
  Interventions: Radiation: Spine Stereotactic Radiosurgery (SSRS)
- High Dose Spine Stereotactic Radiosurgery (Experimental): Participants randomized to this arm will receive Spine Stereotactic Radiosurgery (SSRS) delivered at a higher dose of 20 Gray (Gy) in a single treatment session.
  Interventions: Radiation: Spine Stereotactic Radiosurgery (SSRS)

INTERVENTIONS:
Radiation: Spine Stereotactic Radiosurgery (SSRS) — A non-invasive procedure that uses highly focused, high-energy radiation beams to precisely target metastatic tumors in the spine. The procedure is delivered using advanced techniques like Intensity Modulated Radiotherapy (IMRT) or Volumetric Modulated Arc Therapy (VMAT/RapidArc), which allow the radiation dose to conform tightly to the shape of the tumor. This approach maximizes the dose to the cancer while carefully sparing surrounding healthy tissues, especially the critical spinal cord. The entire course of treatment is delivered in a single session, guided by on-board imaging to ensure sub-millimeter accuracy.

SUMMARY:
The goal of this clinical trial is to learn if a higher dose of Stereotactic Spine Radiosurgery (SSRS), an advanced radiation technique, is better for treating cancer that has spread to the spine (spinal metastases). The study will also learn about the safety of using a higher dose.

The main questions it aims to answer are:

Does a higher radiation dose lead to fewer treatment failures (meaning the tumor growing back or causing serious side effects) one year after treatment? What are the side effects associated with the high dose compared to the standard dose? How does each radiation dose affect a patient's pain and quality of life?

Researchers will randomly assign participants (like a coin toss) to one of two groups to compare the outcomes:

The Standard Dose Group: Will receive a single radiation treatment of 16 Gy. The High Dose Group: Will receive a single, more powerful radiation treatment of 20 Gy.

Participants in this study will:

Receive a single, one-time, highly-focused radiation treatment (SSRS) to the spinal tumor.

Attend regular follow-up visits at the clinic for checkups and imaging scans (like MRI).

Complete questionnaires about their pain levels and quality of life during these visits.

DETAILED DESCRIPTION:
Study Rationale and Background:

Metastatic cancer to the spine is a significant clinical challenge that can lead to severe pain, neurological compromise, and a diminished quality of life. Stereotactic Spine Radiosurgery (SSRS), also known as Stereotactic Ablative Radiotherapy (SABR), has emerged as a paradigm-shifting treatment. This advanced, non-invasive technique allows for the delivery of a single, highly ablative dose of radiation with unprecedented precision, which has shown excellent rates of pain control and tumor response while minimizing dose to the adjacent, critical spinal cord.

Despite the widespread adoption and promising results of SSRS, the optimal dose-fractionation schedule remains an area of active investigation. Previous research, including the landmark RTOG 0631 trial, has established single-fraction 16 Gy as an effective regimen. However, other evidence suggests that a higher radiation dose may lead to more durable local tumor control. This prospective, randomized phase II study, known as the SHINE trial, is designed to formally compare the efficacy and safety of a higher single-fraction dose against the current standard dose.

Study Design and Procedures:

This is a two-arm, parallel-group, randomized, open-label, multi-center study. After providing informed consent and confirming eligibility, participants will be randomly assigned on a 1:1 basis to receive either the standard dose or the high dose of SSRS. The randomization process will incorporate a minimization procedure to ensure balance between the two arms for the key prognostic factor of epidural or paraspinal tumor extension.

The core intervention for all participants is a single session of SSRS. The treatment will be meticulously planned using fused CT and MRI scans to accurately delineate the tumor (Gross Tumor Volume, GTV) and the area at potential microscopic risk (Clinical Target Volume, CTV), following international consensus guidelines from the International Spine Radiosurgery Consortium (ISRC). Radiation will be delivered using state-of-the-art techniques (IMRT or VMAT/RapidArc) with rigorous on-board image guidance to ensure accuracy. Strict dose constraints will be applied to protect the spinal cord and other nearby organs at risk.

Follow-up and Data Collection:

Following treatment, all participants will enter a comprehensive follow-up phase lasting up to two years. The schedule includes regular clinical evaluations, neurological assessments, and serial imaging (MRI and/or CT) to monitor treatment response and detect any potential late toxicities. Additionally, participants will complete validated questionnaires to assess changes in pain and health-related quality of life. Blood samples will be collected at baseline for correlative science studies to investigate potential genetic biomarkers (such as DDR2) and circulating factors that may predict treatment response or risk of skeletal side effects. This robust data collection will allow for a thorough comparison of the two treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologic diagnosis of non-hematopoietic malignancy
2. Radiographic evidence of localized spine metastases without leptomeningeal involvement or intramedullary lesion
3. Maximum four separate sites with a maximal involvement of two continuous vertebral levels
4. Patients do not have prior radiotherapy to the index spine(s)
5. Age ≥ 18 years
6. Karnofsky performance status (KPS) ≥ 60%.
7. Life expectancy ≥ 12 months.
8. Women of childbearing potential and male participants must practice adequate contraception
9. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion Criteria:

1. Prior radiotherapy or radiosurgery to the index spine(s)
2. Serum creatinine > 2.0 mg/dL within 90 days prior registration
3. Contraindication to MR imaging such as implanted metal devices or foreign bodies, severe claustrophobia
4. Patients with metastatict epidural spinal cord compression (≥ grade 2) at the index spine(s) indicative of upfront spine surgery
5. Inability to tolerate treatment procedure
6. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration
   3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   7. Uncontrolled psychiatric disorder
7. Will receive any other investigational agent or chemotherapy and/or target therapies during treatment
8. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic
9. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Composite Treatment Failure at 12 Months | At 12 months after the single fraction of Spine Stereotactic Radiosurgery (SSRS).
  This is a composite endpoint that measures the percentage of participants in each arm who experience a treatment failure. A treatment failure is defined as the first occurrence of either of the following events:
  Clinically Significant Toxicity: The occurrence of a Grade 3 or higher adverse event that is definitely, probably, or possibly related to the radiation treatment. This includes specific neurological, musculoskeletal (e.g., spinal fracture), or gastrointestinal events as defined in the protocol.
  Local Tumor Progression: Unequivocal evidence of tumor growth at the treated spinal site, which is significant enough to warrant further medical intervention, such as spinal surgery or re-irradiation.

SECONDARY OUTCOMES:
Health-Related Quality of Life (EORTC QLQ-C15-PAL) | Baseline, and at 1, 3, 6, 9, and 12 months post-treatment, and then every 3 months for a total follow-up period of up to 24 months.
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Palliative Care (EORTC QLQ-C15-PAL), Taiwan version. This is a 15-item self-reported questionnaire assessing function and symptoms. Scores are converted to a 0-100 scale, with higher functional scores and lower symptom scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: No